CLINICAL TRIAL: NCT02967497
Title: An Open Label Study of UanQiHuoLi Tang Plus Cisplatin-based Chemotherapy in Advanced Epidermal Growth Factor Receptor Wild Type Non-small Cell Lung Cancer
Brief Title: Clinical Study of YQ1 Plus Cisplatin-based Chemotherapy in Advanced NSCLC EGFR Wild Type
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-02-003C
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-07

CONDITIONS: Epithelial Growth Factor Receptor Negative Non-small Cell Lung Cancer
Keywords: Chemotherapy; Herbal medicine; Lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blank (No Intervention): No intervention, just observation.
- YQ1 group (Experimental): Cisplatin-based chemotherapy + YQ1
  Interventions: Drug: YQ1

INTERVENTIONS:
Drug: YQ1 — Oral administered powder
  Other Names: a herbal medicine
  Arms: YQ1 group

SUMMARY:
This randomized pilot phase II trial studies the effect of YQ1, a herbal medicine, with cisplatin-based chemotherapy on gut microbiota and immune response in patients with EGFR/ALK wild type non-small cell lung cancer, stage IIIB-IV.

DETAILED DESCRIPTION:
This randomized pilot phase II trial studies the effect of YQ1, a herbal medicine, with cisplatin-based chemotherapy on gut microbiota and immune response in patients with EGFR/ALK wild type non-small cell lung cancer, stage IIIB-IV. Chinese herbal medicine was known to be beneficial adjuvant or alternative medicine for cancer treatment. However, the mechanism was unknown. This study wants to investigate the effect and mechanism of YQ1, which was proved to improve the antitumor immunity, to inhibit cancer progression, and to prolong overall survival of lung adenocarcinoma in a series of preclinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) that is advanced/metastatic (stage IIIB/IV), EGFR/ALK wild type.
* Subjects who plan to receive cisplatin-based chemotherapy.
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* ECOG performance status >= 3
* WBC =< 4,000 cells/μl, ANC =< 1,500/mcL, Platelets =< 100,000/mcL , Hemoglobin =< 9 g/dL,
* Total bilirubin >= 1.5 x upper limit of normal (ULN), AST >= 1.5x ULN, ALT >= 2.5 x ULN, Creatinine >= 1.5x ULN
* Current uncontrolled cardiac disease such as angina or myocardial infarction, congestive heart failure.
* Chronic or current Inflammatory Bowel Disease, post-surgery of intestine, Lynch syndrome, FAP, Peutz-Jegher.
* History of allergic reactions cisplatin
* Pregnant women are excluded; breastfeeding should be discontinued prior to study entry.
* Received any other clinical trail at the same time.
* Current dementia or other cognitive disorders.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1 year

IPD SHARING:
Plan to Share IPD: No